CLINICAL TRIAL: NCT04029480
Title: A Phase 3, Multicenter, Double-blind, Randomized, Placebo-controlled Clinical Study to Evaluate the Safety and Efficacy of Ertugliflozin (MK-8835/PF-04971729) in Pediatric Participants (Ages 10 to 17 Years, Inclusive) With Type 2 Diabetes Mellitus
Brief Title: Ertugliflozin Type 2 Diabetes Mellitus (T2DM) Pediatric Study (MK-8835/PF-04971729) (MK-8835-059)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-059; PHRR190913-002184 (Registry Identifier: PHRR); 2022-501085-21-00 (Registry Identifier: EU CT); U1111-1279-3984 (Registry Identifier: UTN); MK-8835-059 (Other: MSD); 2017-003455-35 (EudraCT Number)
Record Dates: First submitted 2019-07-11; First posted 2019-07-23 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; Insulin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ertugliflozin 5 mg (Experimental): All participants initially received 5 mg ertugliflozin (ERTU) once daily (QD) and placebo to 15 mg ERTU QD until Week 54 (WK54). At Week 12 (WK12), participants who did not meet the up-titration criteria remained on 5 mg ERTU and placebo to 15 mg ERTU. Participants remained on their background metformin with/without insulin treatment throughout the study.
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Placebo to ertugliflozin 15 mg; Biological: Insulin; Drug: Metformin
- Ertugliflozin 5 mg/5 mg (Experimental): All participants initially received 5 mg ERTU QD and placebo to 15 mg ERTU QD until Week 12. Participants remained on their background metformin with/without insulin treatment throughout the study. Participants who met the up-titration criteria at the WK12 second randomization were re-randomized to remain on 5 mg ERTU and placebo to 15 mg ERTU from WK12 to WK54.
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Placebo to ertugliflozin 15 mg; Biological: Insulin; Drug: Metformin
- Ertugliflozin 5 mg/15 mg (Experimental): All participants initially received 5 mg ERTU QD and placebo to 15 mg ERTU QD until Week 12. Participants remained on their background metformin with/without insulin treatment throughout the study. Participants who met the up-titration criteria at the WK12 second randomization were up-titrated to 15 mg ERTU and placebo to 5 mg ERTU from WK12 to WK54.
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Ertugliflozin 15 mg; Drug: Placebo to ertugliflozin 15 mg; Drug: Placebo to ertugliflozin 5 mg; Biological: Insulin; Drug: Metformin
- Placebo (Placebo Comparator): All participants received matched placebo to 5 mg ERTU and 15 mg ERTU from baseline to WK54. Participants remained on their background metformin with/without insulin treatment throughout the study.
  Interventions: Drug: Placebo to ertugliflozin 15 mg; Drug: Placebo to ertugliflozin 5 mg; Biological: Insulin; Drug: Metformin

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — Ertugliflozin 5 mg, oral, 1 tablet QD
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 5 mg; Ertugliflozin 5 mg/15 mg; Ertugliflozin 5 mg/5 mg
Drug: Ertugliflozin 15 mg — Ertugliflozin 15 mg, oral, 1 tablet QD
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 5 mg/15 mg
Drug: Placebo to ertugliflozin 15 mg — Placebo to ertugliflozin 15 mg, oral, 1 tablet QD
Drug: Placebo to ertugliflozin 5 mg — Placebo to ertugliflozin 5 mg, oral, 1 tablet QD
  Arms: Ertugliflozin 5 mg/15 mg; Placebo
Biological: Insulin — Participants on insulin at screening continued to receive a stable dose of background insulin. The initiation and titration of insulin for rescue therapy was at the discretion of the investigator, based on local/regional/country guidelines.
Drug: Metformin — Participants received stable dose of background metformin.

SUMMARY:
This study evaluated the safety and efficacy of ertugliflozin (MK-8835) in pediatric participants with T2DM on metformin with/without insulin. The primary hypothesis of the study was that the addition of ertugliflozin reduces hemoglobin A1C (HbA1C) more than the addition of placebo after 24 weeks of treatment.

DETAILED DESCRIPTION:
Participants were randomized on Day 1 to the following arms:

* 5 mg ERTU and placebo to 15 mg ERTU (5 mg Ertugliflozin)
* placebo to 5 mg ERTU and placebo to 15 mg ERTU (Placebo)

At Week 12, participants who met the up-titration criteria were re-randomized to the following arms for Weeks 12 to 54:

* 5 mg ERTU and placebo to 15 mg ERTU (5 mg/5 mg Ertugliflozin)
* 15 mg ERTU and placebo to 5 mg ERTU (5 mg/15 mg Ertugliflozin) Participants who did not meet the up-titration criteria remained on 5 mg ERTU and placebo to 15 mg ERTU from Week 12 to Week 54.

The placebo arm continued receiving placebo from Week 12 to Week 54.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Be ≥10 years and ≤17 years of age, when the informed consent is signed
* Has diabetes diagnosed by one of the American Diabetes Association (ADA) criteria.
* Has body mass index (BMI) ≥85th percentile at screening OR participant has a history of being overweight or obese at time of diagnosis of Type 2 diabetes mellitus (T2DM).
* T2DM for ≥2 years, OR T2DM for <2 years and a fasting C-peptide value >0.6 ng/mL at Screening.
* On stable metformin monotherapy (≥1500 mg/day, for ≥8 weeks prior to Screening, OR on a stable metformin dose (≥1500 mg/day, for ≥8 weeks prior to Screening and a stable dose of insulin for ≥8 weeks prior to Screening.
* Contraceptive use by male participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Is a non-sterilized female who is currently not sexually active OR who agrees to abstain from heterosexual activity OR who agrees to start contraception prior to initiating sexual activity and who agrees to use an adequate method of contraception. Contraceptive use by females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Have a family member or adult who, along with the participant, will be closely involved in the participant's daily activities (in the opinion of the investigator) and in the participant's treatment and study procedures.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has known type 1 diabetes mellitus or documented evidence of positive diabetes autoantibodies performed when participant was diagnosed with diabetes.
* Has known monogenic diabetes, or secondary diabetes.
* Has symptomatic hyperglycemia and/or moderate to large ketonuria requiring immediate initiation of another antihyperglycemic agent, including insulin.
* Has a known hypersensitivity or intolerance to any sodium glucose co-transporter 2 (SGLT2) inhibitor.
* Is pregnant, or breast feeding or is expecting to conceive or donate eggs during the study, including 14 days following the last dose of study medication.
* Has previously taken an SGLT2 inhibitor (such as canagliflozin, dapagliflozin, empagliflozin, or ertugliflozin) or was enrolled in a study for these agents.
* Has a history of idiopathic acute pancreatitis or chronic pancreatitis.
* Has a history of severe hypoglycemia while on insulin.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (104):
- United States (11):
  - The University of Alabama at Birmingham ( Site 2207), Birmingham, Alabama
  - Children's Hospital - Los Angeles ( Site 2201), Los Angeles, California
  - Center of Excellence in Diabetes and Endocrinology ( Site 2203), Sacramento, California
  - Memorial Regional Hospital-Joe DiMaggio Children's Hospital Division of Pediatric Endocrinology ( Si, Hollywood, Florida
  - ICCT Research International, Inc. ( Site 2211), Chicago, Illinois
  - Barry J. Reiner MD LLC ( Site 2204), Baltimore, Maryland
  - William Beaumont Hospital ( Site 2219), Royal Oak, Michigan
  - CHEAR Center LLC ( Site 2200), The Bronx, New York
  - Coastal Children''s Services ( Site 2202), Wilmington, North Carolina
  - The Children's Hospital of Philadelphia ( Site 2205), Philadelphia, Pennsylvania
  - Southern Endocrinology and Associates PA ( Site 2218), Mesquite, Texas
- Cliniques Universitaires Saint-Luc ( Site 2300), Brussels, Bruxelles-Capitale, Region de, Belgium
- Canada (2):
  - London Health Sciences Centre ( Site 0002), London, Ontario
  - Hopital Maisonneuve-Rosemont CIUSSS de l Est de L Ile de Montreal ( Site 0001), Montreal, Quebec
- Colombia (2):
  - Centro De Diabetes Cardiovascular IPS Ltda ( Site 0101), Barranquilla, Atlántico
  - MedPlus Medicina Prepagada S.A. ( Site 0102), Bogotá, Bogota D.C.
- Clinica Los Yoses ( Site 0200), San José, Costa Rica
- Hospital Infantil Dr. Robert Reid Cabral ( Site 0300), Santo Domingo, Nacional, Dominican Republic
- France (2):
  - CHU du BOCAGE ( Site 0407), Dijon, Cote-d Or
  - CHU Amiens Hopital Sud ( Site 0413), Amiens, Picardie
- Guatemala (3):
  - Consultorio Privado Dr. Geraldine Utrilla ( Site 0501), Chiquimula
  - Endopedia ( Site 0503), Guatemala City
  - Private Practice - Dr. Flor de Maria Ranchos Monterroso ( Site 0502), Guatemala City
- Hungary (8):
  - Pecsi Tudomanyegyetem Klinikai Kozpont Gyermekgyogyaszati Klinika ( Site 0708), Pécs, Baranya
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház-Gyermekosztály ( Site 0705), Békéscsaba, Bekescsaba
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi OktatoKorhaz ( Site 0701), Miskolc, Borsod-Abauj Zemplen county
  - Vita Verum Medical Egeszsegugyi Szolgaltato Bt ( Site 0706), Székesfehérvár, Fejér
  - Petz Aladar Megyei Oktato Korhaz ( Site 0709), Győr, Győr-Moson-Sopron
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház ( Site 0704), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet ( Site 0702), Budapest
  - Semmelweis Egyetem II. sz. Gyermekgyogyaszati Klinika ( Site 0703), Budapest
- Israel (5):
  - Soroka University Medical Center ( Site 0802), Beersheba
  - Armon M.C ( Site 0803), Haifa
  - Rambam Medical Center ( Site 0801), Haifa
  - Hadassah Mount Scopus ( Site 0800), Jerusalem
  - The Edmond and Lily Safra Children s Hospital ( Site 0804), Ramat Gan
- Italy (6):
  - A.O.Universitaria Meyer ( Site 0901), Florence, Tuscany
  - U.O. di Diabetologia dell'Eta Evolutiva - AUSL 2 ( Site 0904), Caltanissetta
  - IRCCS G. Gaslini ( Site 0900), Genova
  - AOU Federico II di Napoli ( Site 0902), Napoli
  - IRCCS Ospedale Pediatrico Bambino Gesu ( Site 0903), Roma
  - Ospedale Regina Margherita ( Site 0905), Torino
- Malaysia (5):
  - Hospital Universiti Sains Malaysia ( Site 1102), Kubang Kerian, Kelantan
  - Hospital Taiping ( Site 1104), Taiping, Perak
  - Hospital Pulau Pinang. ( Site 1101), George Town, Pulau Pinang
  - Hospital Putrajaya ( Site 1103), Putrajaya, Putrajaya
  - University Malaya Medical Centre ( Site 1100), Kuala Lumpur
- Mauritius (2):
  - Life Nova+ ( Site 1203), Forbach, Pamplemousses District
  - Wellkin Hospital ( Site 1200), Moka
- Mexico (10):
  - Unidad de Investigacion Clinica Cardiometabolica de Occidente ( Site 1007), Guadalajara, Jalisco
  - Centro de Investigacion Medica de Occidente S.C. ( Site 1001), Guadalajara, Jalisco
  - CAIMED Investigación en Salud S.A de C.V ( Site 1008), Mexico City, Mexico City
  - Bio Investigación AMARC, S.C. ( Site 1006), Mexico City, Mexico City
  - Unidad Biomedica Avanzada Monterrey S. A. ( Site 1005), Monterrey, Nuevo León
  - Unidad de Medicina Especializada SMA ( Site 1004), San Juan del Río, Querétaro
  - Consultorio Medico de Endocrinologia Pediatrica ( Site 1002), Culiacán, Sinaloa
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares ( Site 1003), Madero, Tamaulipas
  - Centro de Investigacion Medica Aguascalientes ( Site 1000), Aguascalientes
  - Centro de Atencion e Investigacion Clinica SC ( Site 1009), Aguascalientes
- Philippines (3):
  - Davao Doctors Hospital ( Site 1400), Davao City, Davao Del Sur
  - Institute for Studies on Diabetes Foundation Inc. ( Site 1402), Marikina City, National Capital Region
  - West Visayas State University Medical Center ( Site 1401), Iloilo City
- Poland (4):
  - IN VIVO ( Site 1501), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Poradnia Chorob Metabolicznych. Centrum Zdrowia Tuchow ( Site 1500), Wierzchosławice, Lesser Poland Voivodeship
  - Instytut Diabetologii Sp z o o ( Site 1512), Warsaw, Masovian Voivodeship
  - Clinical Medical Research Sp. z o.o. ( Site 1511), Katowice, Silesian Voivodeship
- Russia (9):
  - Bashkir State Medical University Hospital ( Site 1603), Ufa, Baskortostan, Respublika
  - Federal State Budget Institution Endocrinological Research Center ( Site 1611), Moscow, Moscow
  - Children's City Clinical Hospital #1 ( Site 1604), Novosibirsk, Novosibirsk Oblast
  - Rostov Scientific Research Institution of Obstetrics and Pediatry ( Site 1606), Rostov-on-Don, Rostov Oblast
  - Samara City Pediatric Clinical Hospital n.a. N.N. Ivanova ( Site 1610), Samara, Samara Oblast
  - St.Petersburg State Pediatric Medical University ( Site 1600), Saint Petersburg, Sankt-Peterburg
  - Kazan State Medical University ( Site 1601), Kazan', Tatarstan, Respublika
  - Siberian State Medical University ( Site 1602), Tomsk, Tomsk Oblast
  - Voronezh State Medical University named after N.N.Burdenko ( Site 1608), Voronezh, Voronezskaja Oblast
- Saudi Arabia (7):
  - Hera General Hospital ( Site 1725), Mecca, Al Bahah Region
  - King Abdul Aziz Medical City. National Guard Health Affairs ( Site 1715), Jeddah, Makkah Al Mukarramah
  - King Abdulaziz Medical City - Al Ahsa ( Site 1730), Al Ahsa, Riyadh Region
  - King Abdul Aziz Medical City - AlRiyadh ( Site 1700), Riyadh, Riyadh Region
  - King Abdul Aziz Medical City - AlRiyadh ( Site 1705), Riyadh, Riyadh Region
  - King Salman bin Abdulaziz hospital - Al Riyadh ( Site 1720), Riyadh, Riyadh Region
  - King Salman bin Abdulaziz hospital Al Riyadh ( Site 1710), Riyadh, Riyadh Region
- Turkey (Türkiye) (4):
  - I. U. Cerrahpasa Tip Fakultesi ( Site 2406), Istanbul, Istanbul
  - Cukurova Uni. Tip Fakultesi ( Site 2403), Adana
  - Ankara Bilkent Şehir Hastanesi-Çocuk Hastanesi, Çocuk Endokrinoloji ( Site 2407), Ankara
  - Marmara Üniversitesi Prof. Dr. Asaf Ataseven Hospital ( Site 2400), Istanbul
- Ukraine (9):
  - Chernivtsi Regional Children Clinical Hospital No. 1-Department of Pediatrics and Medical Genetics (, Chernivtsi, Chernivetska Oblast
  - SI Dnipropetrovsk Regional Children Clinical Hospital DOR ( Site 1914), Dnipro, Dnipropetrovsk Oblast
  - MHI Regional Childrens Clinical Hospital ( Site 1908), Kharkiv, Kharkivs’ka Oblast’
  - Institute of Children and Adolescents Health Care of the Academy of Medical Sciences ( Site 1915), Kharkiv, Kharkivs’ka Oblast’
  - Ukr Center of Endocrine Surgery and Transplatation MOH Ukraine ( Site 1903), Kyiv, Kyivska Oblast
  - Medical Center Verum ( Site 1913), Kyiv, Kyivska Oblast
  - Institute of Endocrinology and Metabolism n.a. Komissarenko ( Site 1905), Kyiv, Kyivska Oblast
  - Odessa Regional Children Clinical Hospital ( Site 1912), Odesa, Odesa Oblast
  - Vinnitsa Regional Endocrinology Dispensary, VNMU n.a. M.I.Pyrogov ( Site 1901), Vinnytsia, Vinnytsia Oblast
- United Arab Emirates (6):
  - Dubai Diabetes Center ( Site 2002), Dubai, Dubayy
  - Mustafa Al Qaysi Medical Centre ( Site 2010), Dubai, Dubayy
  - Mediclinic City Hospital ( Site 2005), Dubai, Dubayy
  - Al Jalila Children s Specialty Hospital ( Site 2004), Dubai, Dubayy
  - Thumbay University Hospital ( Site 2001), Ajman
  - Rashid Center For Diabetes and Research ( Site 2006), Ajman
- United Kingdom (3):
  - Royal London Hospital (Whitechapel) ( Site 2100), London, London, City of
  - Chelsea and Westminster Hospital ( Site 2103), London, London, City of
  - West Middlesex University Hospital ( Site 2104), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26199&tenant=MT_MSD_9011
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened up to 4 weeks before dosing. Participants were confirmed at screening to have T2DM for ≥2 years, conform to T2DM protocol specific requirements and be on stable metformin with or without insulin.
  The first randomization was stratified according to the following factors collected at screening: age (10 to 14 years of age/15 to 17 years) and insulin use (yes/no).
  Treatment randomization at Week 12 was stratified according to insulin use (yes/no) at screening.
Groups:
- 5 mg Ertugliflozin: Participants received 5 mg ertugliflozin (ERTU) once daily (QD) and placebo to 15 mg ERTU QD until Week 54 (WK54). At Week 12 (WK12), participants who did not meet the up-titration criteria remained on 5 mg ERTU and placebo to 15 mg ERTU. Participants remained on their background metformin with/without insulin treatment throughout the study.
- 5 mg/5 mg Ertugliflozin: Participants initially received 5 mg ERTU QD and placebo to 15 mg ERTU QD until WK12. Participants remained on their background metformin with/without insulin treatment throughout the study. Participants who met the up-titration criteria at the WK12 second randomization were re-randomized to remain on 5 mg ERTU and placebo to 15 mg ERTU from WK12 to WK54.
- 5 mg/15 mg Ertugliflozin: Participants initially received 5 mg ERTU QD and placebo to 15 mg ERTU QD until WK12. Participants remained on their background metformin with/without insulin treatment throughout the study. Participants who met the up-titration criteria at the WK12 second randomization were up-titrated to 15 mg ERTU and placebo to 5 mg ERTU from WK12 to WK54.
- Placebo: Participants received matched placebo to 5 mg ERTU and 15 mg ERTU from baseline to WK54. Participants remained on their background metformin with/without insulin treatment throughout the study.
Period: Overall Study
Arm/Group | 5 mg Ertugliflozin | 5 mg/5 mg Ertugliflozin | 5 mg/15 mg Ertugliflozin | Placebo
Started | 63 | 22 | 26 | 55
Re-Randomized | 0 (Participants in this arm did not meet the up-titration criteria and were not re-randomized.) | 22 | 26 | 0
Completed | 61 | 22 | 23 | 53
Not Completed | 2 | 0 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Ertugliflozin | 5 mg/5 mg Ertugliflozin | 5 mg/15 mg Ertugliflozin | Placebo | Total
Number analyzed (Participants) | 63 | 22 | 26 | 55 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (2.0) | 14.6 (2.0) | 15.6 (1.8) | 15.1 (1.7) | 14.8 (1.9)
Age, Customized [Count of Participants; unit: Participants] — Per protocol, all participants were randomized before their 18th birthday. Ages from baseline (Day 1) are reported. Participants may show as ≥18 years of age since to protect participant privacy, only the month and year of birth were collected and an imputed date (first of the month) was used to calculate ages in the baseline characteristics; however, each participant was confirmed to be <18 years of age at the time of randomization.
  Participants
    In utero | 0 | 0 | 0 | 0 | 0
    Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0
    Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0
    Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0
    Children (2-11 years) | 6 | 2 | 0 | 1 | 9
    Adolescents (12-17 years) | 56 | 20 | 24 | 52 | 152
    Adults (18-64 years) | 1 | 0 | 2 | 2 | 5
    From 65-84 years | 0 | 0 | 0 | 0 | 0
    85 years and over | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 10 | 20 | 30 | 98
  Male | 25 | 12 | 6 | 25 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 8 | 9 | 22 | 72
  Not Hispanic or Latino | 30 | 13 | 17 | 33 | 93
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 5 | 5 | 19
  Asian | 7 | 5 | 3 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 1 | 5
  White | 43 | 12 | 13 | 31 | 99
  More than one race | 7 | 2 | 1 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline A1C [Mean (Standard Deviation); unit: A1C Percentage] — Hemoglobin A1C is a measure of the percentage of glycated HbA1C in the blood. Participant whole blood samples were collected at baseline to measure A1C. All participants randomized were included in the analysis.
  A1C Percentage | 7.6 (1.0) | 8.5 (1.1) | 8.8 (0.9) | 8.0 (1.0) | 8.0 (1.1)
Insulin Use at Screening [Count of Participants; unit: Participants] — Participant insulin use at screening was assessed. All participants randomized were included in the analysis.
  Participants
    Yes | 18 | 14 | 17 | 24 | 73
    No | 45 | 8 | 9 | 31 | 93
Age at Screening [Number; unit: Years] — The participant age at screening was collected in order to stratify participants at the first randomization.
  Years
    10 to 14 years of age | 27 | 11 | 8 | 23 | 69
    15 to 17 years of age | 36 | 11 | 18 | 32 | 97

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (HbA1C) at Week 24 (Combined Ertugliflozin Versus Placebo)
Description: Hemoglobin A1C is a measure of the percentage of glycated HbA1C in the blood. Participant whole blood samples were collected at baseline and Week 24 to determine the A1C change from baseline (i.e., % A1C at Week 24 minus % A1C at baseline). A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication. The Bayesian mean change from baseline for each combined ertugliflozin and placebo are reported. Per protocol, the ertugliflozin arms are combined for this analysis.
Time Frame: Baseline and Week 24
Population: This analysis includes all participants who received at least 1 dose of study treatment and excludes data following initiation of rescue therapy as well as data collected more than 5 days after the discontinuation of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Groups:
- Combined Ertugliflozin: Participants who received at least 1 dose of ertugliflozin.
Arm/Group | Combined Ertugliflozin | Placebo
Number analyzed (Participants) | 111 | 55
A1C Percentage | -0.55 [-0.82 to -0.28] | 0.12 [-0.23 to 0.47]
Statistical Analysis 1: Comparison: Combined Ertugliflozin vs Placebo; This analysis is based on a Bayesian ANCOVA model including terms for Baseline A1C, treatment, age (10 to 14 years/15 to 17 years), and insulin use (yes/no) at Screening and calculated by Rubin's Rule. The 95% confidence interval actually refers to a credible interval; Test type: Superiority; Difference in Bayesian Means = -0.67, 95% CI 2-sided [-1.06 to -0.29]

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE) Up to Week 24
Description: An adverse event -- Select --is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. Per protocol, the ertugliflozin arms are combined for this analysis.
Time Frame: Up to Week 24
Population: The analysis population includes all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Ertugliflozin | Placebo
Number analyzed (Participants) | 111 | 55
Participants | 59 | 33
Statistical Analysis 1: Comparison: Combined Ertugliflozin vs Placebo; This analysis is based on Miettinen & Nurminen method; Test type: Other; Difference in Percent = -6.8, 95% CI 2-sided [-22.2 to 9.3]

3. Primary Outcome: Number of Participants Who Experienced an AE Up to Week 54
Description: An adverse event is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event. Per protocol, the ertugliflozin arms are combined for this analysis.
Time Frame: Up to Week 54
Population: The analysis population includes all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Ertugliflozin | Placebo
Number analyzed (Participants) | 111 | 55
Participants | 71 | 42
Statistical Analysis 1: Comparison: Combined Ertugliflozin vs Placebo; This analysis is based on Miettinen & Nurminen method; Test type: Other; Difference in Percent = -12.4, 95% CI 2-sided [-25.9 to 2.8]

4. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE Up to Week 24
Description: as for outcome 3
Time Frame: Up to Week 24
Population: The analysis population includes all randomized participants who received at least one dose of study treatment up.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Ertugliflozin | Placebo
Number analyzed (Participants) | 111 | 55
Participants | 0 | 0
Statistical Analysis 1: Comparison: Combined Ertugliflozin vs Placebo; This analysis is based on Miettinen & Nurminen method; Test type: Other; Difference in Percent = 0.00 — No confidence intervals (CIs) were calculated. CIs were computed only for those endpoints where at least ≥8 participants in the combined ertugliflozin group or ≥2 participants in the placebo group had events

5. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE Up to Week 54
Description: as for outcome 3
Time Frame: Up to Week 54
Population: The analysis population includes all randomized participants who received at least one dose of study treatment up.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Ertugliflozin | Placebo
Number analyzed (Participants) | 111 | 55
Participants | 0 | 1
Statistical Analysis 1: Comparison: Combined Ertugliflozin vs Placebo; This analysis is based on Miettinen & Nurminen method; Test type: Other; Difference in Percent = -1.8 — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Change From Baseline in Hemoglobin A1C at Week 24 (Dose-optimized Ertugliflozin Versus Placebo)
Description: Hemoglobin A1C is a measure of the percentage of glycated HbA1C in the blood. Participant whole blood samples were collected at baseline and Week 24 to determine the A1C change from baseline (i.e., % A1C at Week 24 minus % A1C at baseline). A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication.
Time Frame: Baseline and Week 24
Population: This analysis includes all participants who were randomized to ertugliflozin and either did not meet the re-randomization criteria at Week 12 or were re-randomized to ertugliflozin 15 mg, took at least 1 dose of study treatment, and includes all data following initiation of rescue therapy as well as data collected after the discontinuation of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Groups:
- Dose-Optimized Ertugliflozin: Participants who were randomized to ertugliflozin and either did not meet the re-randomization criterion at Week 12 or were re-randomized to 15 mg ertugliflozin.
Arm/Group | Dose-Optimized Ertugliflozin | Placebo
Number analyzed (Participants) | 89 | 55
A1C Percentage | -0.42 [-0.76 to -0.08] | 0.25 [-0.22 to 0.72]
Statistical Analysis 1: Comparison: Dose-Optimized Ertugliflozin vs Placebo; This analysis is based on an ANCOVA model including terms for Baseline A1C, treatment, age (10 to 14 years/15 to 17 years), and insulin use (yes/no) at Screening and calculated by Rubin's Rule; Test type: Superiority; p = 0.021, ANCOVA; Difference in Least Squares Means = -0.66, 95% CI 2-sided [-1.23 to -0.10]

7. Secondary Outcome: Change From Baseline in Hemoglobin A1C at Week 24 (5 mg Ertugliflozin Versus Placebo)
Description: as for outcome 6
Time Frame: Baseline and Week 24
Population: This analysis includes all participants randomized to ertugliflozin and either did not meet the re-randomization criteria at Week 12 or were re-randomized to 5 mg ertugliflozin, and all data following initiation of rescue therapy as well as data collected after the discontinuation of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: A1C Percentage
Groups:
- 5 mg Ertuglifozin: Participants who were randomized to ertugliflozin and either did not meet the re-randomization criterion at Week 12 or were re-randomized to 5 mg ertugliflozin.
Arm/Group | 5 mg Ertuglifozin | Placebo
Number analyzed (Participants) | 85 | 55
A1C Percentage | -0.54 [-0.86 to -0.22] | 0.32 [-0.11 to 0.76]
Statistical Analysis 1: Comparison: 5 mg Ertuglifozin vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.001, ANCOVA; Difference in Least Squares Means = -0.86, 95% CI 2-sided [-1.39 to -0.33]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Blood glucose is measured on a fasting basis. FPG is expressed as mg/dL. Blood was drawn at predose on Day 1 and after 24 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 24 minus FPG at baseline). A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication. Per protocol, the ertugliflozin arms were combined for this analysis.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Combined Ertugliflozin | Placebo
Number analyzed (Participants) | 111 | 55
mg/dL | -20.8 [-30.8 to -10.8] | 8.2 [-5.4 to 21.7]
Statistical Analysis 1: Comparison: Combined Ertugliflozin vs Placebo; This analysis is based on a constrained longitudinal data analysis (cLDA) model including terms for treatment, time, age (10 to 14 years/15 to 17 years), insulin use (yes/no), interaction of time by treatment with the constraint that the model estimated a single baseline mean (applicable to all treatment groups); Test type: Superiority; p = 0.001, cLDA; Difference in Least Squares Means = -29.0, 95% CI 2-sided [-44.4 to -13.6]

9. Secondary Outcome: Change From Baseline in Hemoglobin A1C at Week 54
Description: Hemoglobin A1C is a measure of the percentage of glycated HbA1C in the blood. Participant whole blood samples were collected at baseline and Week 54 to determine the A1C change from baseline (i.e., A1C at Week 54 minus A1C at baseline). A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received glycemic rescue medication. Per protocol, the ertugliflozin arms were combined for this analysis.
Time Frame: Baseline and Week 54
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: AIC Percentage
Arm/Group | Combined Ertugliflozin | Placebo
Number analyzed (Participants) | 111 | 55
AIC Percentage | -0.22 [-0.59 to 0.16] | 0.81 [0.24 to 1.38]
Statistical Analysis 1: Comparison: Combined Ertugliflozin vs Placebo; This analysis is a based on a constrained longitudinal data analysis (cLDA) model including terms for treatment, time, age (10 to 14 years/15 to 17 years), insulin use (yes/no), interaction of time by treatment with the constraint that the model estimated a single baseline mean (applicable to all treatment groups); Test type: Superiority; p = 0.003, cLDA; Difference in Least Squares Means = -1.03, 95% CI 2-sided [-1.70 to -0.35]

10. Secondary Outcome: Change From Baseline in FPG at Week 54
Description: Blood glucose is measured on a fasting basis. FPG is expressed as mg/dL. Blood was drawn at predose on Day 1 and after 54 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 54 minus FPG at baseline). A negative number indicates a reduction in FPG. Participants who met glycemic rescue criteria received glycemic rescue medication. Per protocol, the ertugliflozin arms were combined for this analysis.
Time Frame: Baseline and Week 54
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Combined Ertugliflozin | Placebo
Number analyzed (Participants) | 111 | 55
mg/dL | -12.1 [-23.7 to -0.5] | 21.0 [3.6 to 38.4]
Statistical Analysis 1: Comparison: Combined Ertugliflozin vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.001, cLDA; Difference in Least Squares Means = -33.1, 95% CI 2-sided [-53.0 to -13.1]

ADVERSE EVENTS:
Time Frame: Up to 56 weeks.
Description: All-Cause Mortality is reported for all randomized participants. Serious adverse events and other adverse events are reported for all participants who received at least 1 dose of treatment.
Groups:
- 5 mg Ertugliflozin: Week 1-54: Participants received 5 mg ertugliflozin (ERTU) once daily (QD) and placebo to 15 mg ERTU QD until Week 54 (WK54). At Week 12 (WK12), participants who did not meet the up-titration criteria remained on 5 mg ERTU and placebo to 15 mg ERTU. Participants remained on their background metformin with/without insulin treatment throughout the study.
- 5 mg/5 mg Ertugliflozin: Week 1-54: Participants initially received 5 mg ERTU QD and placebo to 15 mg ERTU QD until WK12. Participants remained on their background metformin with/without insulin treatment throughout the study. Participants who met the up-titration criteria at the WK12 second randomization were re-randomized to remain on 5 mg ERTU and placebo to 15 mg ERTU from WK12 to WK54.
- 5 mg/15 mg Ertugliflozin: Week 1-12 (Ertu 5 mg): After the first randomization on Day 1, participants received 5mg ERTU QD and placebo to 15 mg ERTU QD until WK12. Participants remained on their background metformin with/without insulin treatment throughout the study.
- 5 mg/15 mg Ertugliflozin: Week 12-54 (Ertu 15 mg): After the second randomization at WK12, participants received 15mg ERTU QD and placebo to 5 mg ERTU QD from WK12 to WK54. Participants remained on their background metformin with/without insulin treatment throughout the study.
- Placebo: Week 1-54: Participants received matched placebo to 5 mg ERTU and 15 mg ERTU from baseline to WK54. Participants remained on their background metformin with/without insulin treatment throughout the study.
Arm/Group | 5 mg Ertugliflozin: Week 1-54 | 5 mg/5 mg Ertugliflozin: Week 1-54 | 5 mg/15 mg Ertugliflozin: Week 1-12 (Ertu 5 mg) | 5 mg/15 mg Ertugliflozin: Week 12-54 (Ertu 15 mg) | Placebo: Week 1-54
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/22 | 0/26 | 0/26 | 0/55
Serious Adverse Events (participants affected / at risk) | 2/63 | 1/22 | 0/26 | 1/26 | 0/55
Other Adverse Events (participants affected / at risk) | 29/63 | 11/22 | 8/26 | 14/26 | 31/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Ertugliflozin: Week 1-54 (N=63) | 5 mg/5 mg Ertugliflozin: Week 1-54 (N=22) | 5 mg/15 mg Ertugliflozin: Week 1-12 (Ertu 5 mg) (N=26) | 5 mg/15 mg Ertugliflozin: Week 12-54 (Ertu 15 mg) (N=26) | Placebo: Week 1-54 (N=55)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Ertugliflozin: Week 1-54 (N=63) | 5 mg/5 mg Ertugliflozin: Week 1-54 (N=22) | 5 mg/15 mg Ertugliflozin: Week 1-12 (Ertu 5 mg) (N=26) | 5 mg/15 mg Ertugliflozin: Week 12-54 (Ertu 15 mg) (N=26) | Placebo: Week 1-54 (N=55)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 4 (4)
Gastritis (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (2) | 2 (2) | 4 (4) | 3 (3)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 1 (2) | 0 (0) | 2 (2) | 4 (4)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Influenza (Infections and infestations) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 5 (6) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 1 (1) | 1 (1) | 1 (1) | 6 (8)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (35) | 2 (3) | 3 (12) | 5 (40) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1) | 3 (4) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT04029480/Prot_SAP_000.pdf